CLINICAL TRIAL: NCT04963205
Title: Sleep Position and Sleep Quality in Chronic Obstructive Pulmonary Disease- a Prospective, Open Label, Randomized, Cross-over Clinical Trial
Brief Title: Sleeping Position Study in COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lowie Vanfleteren (Other Government)
Responsible Party: Sponsor-Investigator, Lowie Vanfleteren, Principal Investigator, Head of COPD-center, Vastra Gotaland Region
Organization: Vastra Gotaland Region (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Sovposition studie
Record Dates: First submitted 2021-06-08; First posted 2021-07-15 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: COPD; Sleep
Keywords: COPD; Sleep; Sleep positions; Adjustable bed backrest
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjustable bed backrest (Experimental): Sleeping in elevated body position (>30 degrees from supine position) for 4 weeks is a requirement for the intervention group. Patients can define their own most comfortable position during the night.
  Interventions: Device: Adjustable bed backrest
- Usual bed (Active Comparator): Sleeping in a standard bed and "flat" (<30 degrees from supine position) position for 4 weeks. Patients can define their own most comfortable position during the night.
  Interventions: Other: Standard bed

INTERVENTIONS:
Device: Adjustable bed backrest — The adjustable bed backrest facilitates for the individual high lying with a fowler (90 degrees raised head and trunk) and/or semi fowler position (30-45 degrees raised head and trunk) which enables patient's lung expansion. The diaphragm is pulled downwards by the gravity allowing for lung expansion and improved ventilation. In addition, the upper airways are stretched in order to prevent upper airway narrowing during sleep (flow limitation, snoring, obstructive sleep apnea). The position relaxes the tension of the abdominal muscles, allowing for improved breathing. Patients can define their own most comfortable position during the night. Elevated body position over 30 degrees from supine position is a requirement for the intervention group. No sleeping time restrictions will be applied. One week washout period between the interventions will be used.
  Arms: Adjustable bed backrest
Other: Standard bed — Sleeping in a standard bed, in a position below 30 degrees from supine position. No sleeping time restrictions will be applied. One week washout period between the interventions will be used.
  Arms: Usual bed

SUMMARY:
Background: Chronic obstructive pulmonary disease (COPD) is a common chronic disease characterized by persistent respiratory symptoms and airflow restriction, due to airway and/ or alveolar abnormalities usually caused by significant exposure to harmful particles or gases, in particular cigarette smoking. Sleep disorders are common in society and it is not surprising that they also affect individuals with COPD. Patients with COPD, especially those in severe stages of the disease suffer from many sleep disorders and its prevalence varies depending on the disease. Epidemiological studies report that approximately 75% of COPD patients experience nocturnal symptoms of the disease. The most common are sleep-breathing disorders (nocturnal hypoxemia, central sleep apnea, difficulty breathing, sleep-related hypoventilation), insomnia and sensory motor disorders during sleep, including restless legs syndrome. Patients with COPD not only experience poorer sleep quality and concomitant sleep disorders but also have a higher chance of sudden nocturnal death, especially during a period of COPD exacerbation.

Scientific studies show that elevated posture during sleep (>30 degrees raised head and back from the supine position) has a positive effect on sleep quality. To date, this has not been proven in patients with COPD who are a special group with sleep disorders.

Research questions and objectives: The primary study objective is to evaluate if adjusted sleeping position with electrical bed backrest improves the quality of sleep in patients with COPD.

The exploratory objectives are:

1. To evaluate if adjusted sleeping position improves total sleep time, respiratory patterns, oxygen saturation and heart rate (measured by CASIS, WatchPat and Sleepiz).
2. To investigate if adjusted sleeping position decreases COPD-related symptoms during sleep and daytime (measured with CAT score).
3. To evaluate if adjusted sleeping position reduces patient's fatigue during the day (measured with FSS questionnaire).
4. To evaluate if better sleep at night is associated with more energy, more activity and less breaks for rest during the day (measured with OQ-S, 6MWT and smartwatch).
5. To compare the results from the two sleep recording technologies (single night minimal contact sleep recorder-WatchPat versus several nights without contact sleep recorder-Sleepiz).

Study design: Prospective, open label, cross-over clinical trial with randomized treatment order. Every subject will use the assigned intervention for 4 weeks. The intervention is an electrical bed backrest used during sleep time. The randomization will be non-adjusted, in ratio 1:1. A total of 40 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed COPD diagnosis
2. FEV1< 50%
3. COPD grade B, D
4. Male or female patients, aged ≥40 years
5. Difficulties with sleep, as defined by result of 4-5 points in sleep-related question in CAT questionnaire
6. A bed that is possible to adjust to the electric bed backrest
7. Signed informed consent form.

Exclusion Criteria:

1. Previous diagnosis or treatment of clinically significant sleep disorder including sleep apnea treated with continuous positive airway pressure (CPAP), insomnia, restless legs syndrome or frequent parasomnia
2. Long-term stay (>1 week) away from home during the study period, where there is no possibility to use the electrical bed backrest.
3. Person that cannot communicate in Swedish language.
4. Unable to comply with study procedures as in the opinion of the study investigator (e.g. other severe diseases with short life expectancy or which make it impossible for the patients to participate in the study, evidence of alcohol or drug abuse, dementia, severe psychiatric disorder)
5. Already enrolled in other studies perceived to interfere with this protocol
6. Clinically significant disorders not allowing to maintain a sitting position during sleep including severe back pain, lumbalgia, spinal stenosis
7. Patients inability or unwillingness to sleep in the sitting position.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Impact of COPD on sleep quality | Baseline, 4 weeks and 9 weeks after baseline
  Change in quality of sleep with be objectively measured by the COPD and Asthma Sleep Impact Scale (CASIS). The 7 question survey, each item scores from 1 to 5 (higher score indicates greater impact) for a maximum of 35. CASIS raw scores can be linearly transformed to a 0-100 total scale score.

SECONDARY OUTCOMES:
Total sleep time | Constant monitoring during 4 weeks of intervention and 4 weeks of control arm for Sleepiz; Baseline, 3 weeks after and 7 weeks after for WatchPAT
  Change in total sleep time will be collected by a WatchPAT device (wrist-mounted device that records PAT signals) and Sleepiz device (contactless device).
Respiratory disturbance index | Baseline, 3 weeks after and 7 weeks after.
  Change in respiratory indices, the respiratory disturbance index (pRDI) will be measured by WatchPAT device.
Number of apneas or hypopneas | Constant monitoring during 4 weeks of intervention and 4 weeks of control arm for Sleepiz; Baseline, 3 weeks after and 7 weeks after for WatchPAT
  Change in respiratory indices, the number of apneas or hypopneas recorded during the study per hour of sleep (pAHI) will be measured by WatchPAT and Sleepiz device.
Oxygen desaturation index | Baseline, 3 weeks after and 7 weeks after.
  Change in the oxygen desaturation index (ODI) will be measured by WatchPAT device.
Oxygen saturation | Baseline, 3 weeks after and 7 weeks after.
  Change in mean oxygen saturation (%) will be measured by WatchPAT device.
Central apnea-hypopnea index | Baseline, 3 weeks after and 7 weeks after.
  Change in respiratory indices, the central apnea-hypopnea index (pAHIc) will be measured by WatchPAT device.
Cheyne-Stokes respiration | Baseline, 3 weeks after and 7 weeks after.
  Change in respiratory indices, the Cheyne-Stokes respiration (%CSR) will be measured by WatchPAT device.
Pulse rate | Constant monitoring during 4 weeks of intervention and 4 weeks of control arm for Sleepiz; Baseline, 3 weeks after and 7 weeks after for WatchPAT
  Change in pulse rate during sleep will be measured by WatchPAT and Sleepiz device
Wake/ sleep stages | Constant monitoring during 4 weeks of intervention and 4 weeks of control arm for Sleepiz; Baseline, 3 weeks after and 7 weeks after for WatchPAT
  Changes in wake/ sleep stages will be measured by WatchPAT and Sleepiz device.
Rapid eye movement stage time | Baseline, 3 weeks after and 7 weeks after.
  Change in rapid eye movement (REM) phase (%) will be measured by WatchPAT device.
Sleeping body position | Baseline, 3 weeks after and 7 weeks after.
  Change in body position during sleep (supine, non-supine, prone, right, left) will be measured by WatchPAT device.
Breathing rate | Constant monitoring during 4 weeks intervention and 4 weeks control arm.
  Changes in breathing rate (times/minute) will be measured by Sleepiz device.
Respiratory Irregularity Index | Constant monitoring during 4 weeks intervention and 4 weeks control arm.
  Changes in respiratory regularity index will be measured by Sleepiz device.
Snoring level | Baseline, 3 weeks after and 7 weeks after.
  Changes in snoring level (dB) during sleep will be measured by WatchPAT device.
Time in bed | Constant monitoring during 4 weeks intervention and 4 weeks control arm.
  Changes in total time spend in bed (measured in hours and minutes) will be measured by Sleepiz device.
COPD-related symptoms | Baseline, 4 weeks and 9 weeks after baseline
  Change in disease-specific related symptoms will be measured by using a COPD Assessment Test (CAT) questionnaire. CAT measures COPD symptoms with scores from 0 to 5 points (0 indicating no impact or symptoms, 5- worst possible impact or symptoms) summing up to a total CAT score range of 0-40 points.
Fatigue | Baseline, 4 weeks and 9 weeks after baseline
  Changes in fatigue will be objectively measured by using the Fatigue Severity Scale (FSS). It is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Answers can be scored from 1 to 7 and higher score means greater fatigue severity.
Occupational activity | Baseline, 4 weeks and 9 weeks after baseline
  Changes in occupational questionaire will be objectively measured by using the Occupational Questionnaire, Swedish version (OQ-S). Users classify the activity as work, play or leisure and record their perception of competence, value, and enjoyment for each activity and mark its competence and importance. The OQ-S register time use based on a pre-defined 19-hour window, from 05:00 to 00:00. Using 5-point likert-type scale indicating how well they do the activity, how important is the activity and how enjoyable it is. The higher the score, the better the individual's satisfaction, value and enjoyment of the activity.

CONTACTS AND LOCATIONS:
Locations (1):
- COPD-center, Sahlgrenska University Hospital, Gothenburg, VGR, Sweden